CLINICAL TRIAL: NCT00764049
Title: Prospective Pilot Study Assessing Safety and Efficacy of Single Pass Albumin Dialysis in Patients With Acute on Chronic Liver Failure
Brief Title: Single Pass Albumin Dialysis in Patients With Cirrhosis
Acronym: DACAR
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Laboratoire français de Fractionnement et de Biotechnologies (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P050902
Record Dates: First submitted 2008-09-30; First posted 2008-10-01 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Cirrhosis; Acute on Chronic Hepatic Failure; Hepatorenal Syndrome; Encephalopathy
Keywords: Albumin dialysis; Artificial liver support; Acute on chronic liver failure
MeSH Terms: conditions — Fibrosis; Hepatorenal Syndrome; Brain Diseases; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1: Single pass albumin dialysis (Experimental): Patients entered in the pilot study.
  Interventions: Device: Single pass albumin dialysis

INTERVENTIONS:
Device: Single pass albumin dialysis — 6 hours sessions of albumin dialysis.

SUMMARY:
The aim of this study is to determine whether a simplified device of albumin dialysis also has beneficial effects.

DETAILED DESCRIPTION:
Albumin dialysis has beneficial effects in patients with acute on chronic liver failure. However, current devices are complex and costly. The aim of this study is to determine whether a simplified device of albumin dialysis also has beneficial effects.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Written consent after information of the patient or, in case of inability, by a parent or a close if he is present.
* Patient having a cirrhosis researched by previous exams (liver biopsy) or, in the absence of previous diagnosis, diagnosed in view of the results of clinical, biological and morphological data, whatever the origin of the cirrhosis (virus of hepatitis B, virus of hepatitis C, extreme consumption of alcohol or other reasons)

Exclusion Criteria:

* Participation to an other study in the 4 weeks before
* Active digestive bleeding, unchecked by the pharmacological treatments and the endoscopic techniques.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-06; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Effects on clinical and biochemical variables | 3 months follow-up

SECONDARY OUTCOMES:
Safety | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: François Durand, Pr, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France